CLINICAL TRIAL: NCT03887936
Title: Testosterone Therapy and Bone Quality in Men With Diabetes and Hypogonadism
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDB-009-18F; 1I01CX001665-01A2 (NIH)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus; Hypogonadism
Keywords: diabetes mellitus; hypogonadism; testosterone; bone quality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism; Diabetes Mellitus | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled study comparing the effect of testosterone therapy in men with both type 2 diabetes mellitus and hypogonadism on bone quality, bone turnover markers and circulating osteoblast and osteoclast progenitors.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: No other parties will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Testosterone arm (Experimental): Testosterone gel 1.62%
  Interventions: Drug: Testosterone gel 1.62%
- Placebo arm (Placebo Comparator): Matching placebo will be prepared by the Michael DeBakey VA Medical Center Pharmacy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone gel 1.62% — Testosterone gel 1.62%, apply 2 pumps to upper arm and shoulder.
  Other Names: Androgel
  Arms: Testosterone arm
Drug: Placebo — Matching placebo gel, apply 2 pumps to upper arm and shoulder
  Arms: Placebo arm

SUMMARY:
Low testosterone and diabetes mellitus are each associated with increased risk for fractures. Men with diabetes mellitus are commonly found to have low testosterone as well. Testosterone has been shown to improve the bone health of patients with low testosterone but has not been tested in patients who also have diabetes mellitus in addition to low testosterone. To date, there is no treatment that is specifically recommended for bone disease among patients with diabetes. This study will evaluate the effect of testosterone on the bone health of male Veterans who have both diabetes and low testosterone, both of which are highly prevalent in this subset of the population.

DETAILED DESCRIPTION:
An existing mutual influence between testosterone (T) and glucose metabolism has been suggested by studies showing that men with low T have impaired glucose tolerance, while a significant number of men with type 2 diabetes mellitus (T2D) and obesity have low T. Thus, it is not surprising that as much as 64% of men with T2D were found to have low T. Hypogonadism and diabetes mellitus (DM) each is associated with increased risk for fractures. While hypogonadism is associated with increased bone turnover and bone loss. DM is associated with low bone turnover and normal or high bone mineral density (BMD) but paradoxically a high risk for fractures. The preliminary data showed that compared to non-diabetic hypogonadal men, men with both conditions have suppressed bone turnover, higher volumetric BMD (vBMD) and smaller bone size. As the effect of T on the male skeleton is mainly mediated by its conversion to estradiol (E2) by the enzyme aromatase, the possibility of further suppression of bone turnover with T therapy in these patients would be a concern. However, the investigators' initial data also showed that T therapy in men with both conditions resulted in increased in markers of bone turnover and bone size compared to the decrease in bone turnover and decrease in bone size in men with hypogonadism only, suggesting activation in bone remodeling and improvement in bone geometry in the former. Furthermore, the investigators also found a trend for increase in bone strength (by finite element analysis or FEA) in the limited number of men with both low T and T2D randomized to T compared to placebo. These findings only suggest but do not prove with certainty that T therapy would be beneficial to men with both low T and T2D. The central hypothesis of this study is that T therapy will result in improvement in bone quality in patients who have both hypogonadism and T2D. Thus, the specific aims of this proposal are: 1) to determine the effect of T therapy on bone strength as assessed by finite element analysis ( FEA) using high-resolution peripheral quantitative computer tomography (HR-pQCT), 2) to determine the effect of T therapy on markers of bone turnover, and 3) an exploratory aim, to evaluate the mechanism for improvement in bone quality from T therapy. The investigators hypothesize that because T stimulates osteoblastic proliferation and differentiation, the ensuing increase in osteoblast number will lead to an enhanced cross-talk between osteoblast and osteoclast resulting in activation of bone remodeling and replacement of old with new bone, hence, improvement in bone quality. In this study the investigators will enroll 166 men with T2D and hypogonadism and randomize them to either testosterone gel 1.62% or placebo for 12 months.

The following main outcomes will be evaluated: aim# 1) change in the primary endpoint which is FEA, by HRpQCT, #2) changes in C-telopeptide (CTX) a marker of bone resorption, and aim #3) changes in circulating osteoblast progenitor (COP). The investigators anticipate an increase in FEA at the tibia and radius suggesting improvement in bone strength, increase CTX and increase in circulating osteoblast progenitors. The investigators further anticipate an increase in other markers of bone turnover (both bone formation and resorption) and osteoclast precursors in men with hypogonadism and T2D randomized to T compared to placebo. Given the suppressed bone turnover at baseline in men with low T and T2D, the investigators hypothesize that the beneficial effect of T is its effect in activating bone remodeling ultimately resulting in improvement in bone quality.

Results from this study will provide information on the utility of T not only in improving quality of life but also in improving bone quality in hypogonadal men with T2D. Given the relationship between glucose metabolism and testosterone production, and the increasing number of male patients diagnosed with both hypogonadism and T2D, this study will benefit not only the significant number of male Veterans who have both conditions but also men in general.

ELIGIBILITY:
Inclusion Criteria:

* Male veterans only
* 35 to 70 years old
* With an average fasting morning T level from 2 measurements of <300 ng/dl taken at least a day apart

  * symptoms of hypogonadism as assessed using the androgen deficiency in aging male (ADAM) questionnaire
* Participants should have

  * T2D
  * an A1C of <11.5 %
  * a fasting blood sugar of 180 mg/dl
  * body mass index (BMI) <40 kg/m2
  * with DM of 15 years duration or less to target men who have relatively less complications from long-term DM

Exclusion Criteria:

* history of prostate or breast cancer
* history of testicular disease
* untreated severe sleep apnea
* ongoing illness that could prevent the subject from completing the study
* a hematocrit of >50%
* prostate-related findings as:

  * a palpable prostate nodule on digital rectal exam (DRE)
* serum PSA of 4.0 ng/ml
* International Prostate Symptom Score (IPSS) >19 (severe)
* on androgen therapy or selective androgen receptor modulators
* on medications that affect bone metabolism such as:

  * estrogen
  * selective estrogen receptor modulator as:

    * raloxifene
    * aromatase inhibitors
    * GnRH analogs
    * glucocorticoids with prednisone equivalent of least 5 mg daily for 1 month
    * anabolic steroids
    * phenobarbital and Dilantin
* use of bisphosphonates within two years of study entry, i.e.:

  * risedronate
  * alendronate
  * zoledronic acid
  * pamidronate
* diseases that interfere with bone metabolism, as:

  * hyperparathyroidism
  * untreated hyperthyroidism
  * osteomalacia
  * chronic liver disease
  * renal failure with estimated glomerular filtration rate of <45 ml/min
  * hypercortisolism
  * malabsorption
  * immobilization
* current alcohol use of > 3 drinks/day
* those with a history of:

  * deep vein thrombosis
  * pulmonary embolism
  * recent stroke or recent diagnosis of coronary artery disease of < 6 months
* because of the potential of being randomized to placebo, subjects with osteoporosis or a BMD T-score by DXA of -2.5 in the lumbar spine, total femur or femoral neck and those with a history of fragility fractures

  * spine
  * hip
  * wrist

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Reina C. Villareal, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russo V, Chen R, Armamento-Villareal R. Hypogonadism, Type-2 Diabetes Mellitus, and Bone Health: A Narrative Review. Front Endocrinol (Lausanne). 2021 Jan 18;11:607240. doi: 10.3389/fendo.2020.607240. eCollection 2020. PMID 33537005
- [Background] Deepika F, Ballato E, Colleluori G, Aguirre L, Chen R, Qualls C, Villareal DT, Armamento-Villareal R. Baseline Testosterone Predicts Body Composition and Metabolic Response to Testosterone Therapy. Front Endocrinol (Lausanne). 2022 Jul 11;13:915309. doi: 10.3389/fendo.2022.915309. eCollection 2022. PMID 35898448
- [Background] Bathina S, Armamento-Villareal R. The complex pathophysiology of bone fragility in obesity and type 2 diabetes mellitus: therapeutic targets to promote osteogenesis. Front Endocrinol (Lausanne). 2023 Jul 20;14:1168687. doi: 10.3389/fendo.2023.1168687. eCollection 2023. PMID 37576965
- [Background] Deepika F, Bathina S, Armamento-Villareal R. Novel Adipokines and Their Role in Bone Metabolism: A Narrative Review. Biomedicines. 2023 Feb 20;11(2):644. doi: 10.3390/biomedicines11020644. PMID 36831180
- [Background] Bathina S, Prado M, Fuenmayor Lopez V, Colleluori G, Aguirre L, Chen R, Villareal DT, Armamento-Villareal R. PRDM16 Enhances Osteoblastogenic RUNX2 via Canonical WNT10b/beta-CATENIN Pathway in Testosterone-Treated Hypogonadal Men. Biomolecules. 2025 Jan 8;15(1):79. doi: 10.3390/biom15010079. PMID 39858473
- [Background] Chen R, Armamento-Villareal R. Obesity and Skeletal Fragility. J Clin Endocrinol Metab. 2024 Jan 18;109(2):e466-e477. doi: 10.1210/clinem/dgad415. PMID 37440585
- [Result] Russo V, Colleluori G, Chen R, Mediwala S, Qualls C, Liebschner M, Villareal DT, Armamento-Villareal R. Testosterone therapy and bone quality in men with diabetes and hypogonadism: Study design and protocol. Contemp Clin Trials Commun. 2021 Jan 20;21:100723. doi: 10.1016/j.conctc.2021.100723. eCollection 2021 Mar. PMID 33718653
- [Result] Ballato E, Deepika FNU, Russo V, Fleires-Gutierrez A, Colleluori G, Fuenmayor V, Chen R, Villareal DT, Qualls C, Armamento-Villareal R. One-Year Mean A1c of > 7% is Associated with Poor Bone Microarchitecture and Strength in Men with Type 2 Diabetes Mellitus. Calcif Tissue Int. 2022 Sep;111(3):267-278. doi: 10.1007/s00223-022-00993-x. Epub 2022 Jun 4. PMID 35665818
- [Result] Bathina S, Lopez VF, Prado M, Ballato E, Colleluori G, Tetlay M, Villareal DT, Mediwala S, Chen R, Qualls C, Armamento-Villareal R. Health implications of racial differences in serum growth differentiation factor levels among men with obesity. Physiol Rep. 2024 Dec;12(23):e70124. doi: 10.14814/phy2.70124. PMID 39668628
- [Result] Ballato E, Deepika F, Prado M, Russo V, Fuenmayor V, Bathina S, Villareal DT, Qualls C, Armamento-Villareal R. Circulating osteogenic progenitors and osteoclast precursors are associated with long-term glycemic control, sex steroids, and visceral adipose tissue in men with type 2 diabetes mellitus. Front Endocrinol (Lausanne). 2022 Sep 12;13:936159. doi: 10.3389/fendo.2022.936159. eCollection 2022. PMID 36171900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by flyers and letters from the Primary Care and Endocrine Clinics at the Michael E. DeBakey VA Medical Center. The study was open to enrollment on October 1, 2019 and closed on September 30, 2024.
Pre-assignment Details: There were 467 subjects who responded to our study advertisement. Three hundred ninety-five came for orientation, consent and screening, while 72 declined to come. Three hundred three were not enrolled; 271 failed our screening procedures from either laboratory tests or significant past medical history that constitutes an exclusion from the study, 21 did not finish the required screening tests and 11 decided not to proceed with the study.
Period: Overall Study
Arm/Group | Testosterone Arm | Placebo Arm
Started | 46 | 46
Bone Quality Assessments | 34 | 34
Completed | 44 | 42
Not Completed | 2 | 4
Not completed — Relocation | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Arm | Placebo Arm | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 45 | 91
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (6.8) | 55.5 (6.6) | 54.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 46 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 40 | 37 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 24 | 30 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Finite Element Analysis of Bone to Measure Bone Strength
Description: The FEA (or FEA) is a surrogate measure of strength using computational biomechanical principles and integrate bone morphology and bone mass to calculate bone strength under various loading conditions normally seen in daily living activities. In addition, the ratio of load to strength can be calculated by using patient information (i.e. weight and height) and FEA derived bone strength to mechanistically simulate bone failure and thus, whether fracture is likely during a given activity. Using high-resolution peripheral quantitative computer tomography (HRPQCT) we will compute for FEA, using FEA software with images generated using Image Processing Language to estimate the biomechanical properties of the bone. Each bone voxel will be converted to hexahedral finite elements with linear-elastic and isotropic material behavior. The FEA model will be subject to uniaxial compression and stiffness and failure load will be estimated. FEA will be assessed at months 0, 6 and 12.
Time Frame: months 0, 6 and 12
Population: There were 2 dropouts in the testosterone group thus, 44 participants finished the study. However, the imaging studies of one patient who finished the study is not optimum for FEA.
  There were 4 dropouts in the placebo thus, 42 participants finished the study. However, the investigators were unable to assess the finite element analysis in one patient as HRPQCT machine broke down when the participant came for final visit and refused to come again just for this assessment.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Testosterone Arm | Placebo Arm
Number analyzed (Participants) | 43 | 41
% change
  Change (%) from baseline in stiffness of radius at 6 months | 1.2 (8.7) | 1.6 (11.6)
  Change (%) from baseline in failure load of radius at 6 months | 1.6 (10.4) | 0.88 (8.4)
  Change (%) from baseline in stiffness of tibia at 6 months | -0.50 (5.2) | -0.45 (6.8)
  Change (%) from baseline in failure load of tibia at 6 months | -0.41 (8.3) | -0.36 (5.8)
  Change (%) from baseline in stiffness of the radius at 12 months | 0.69 (8.3) | 0.52 (7.5)
  Change (%) from baseline in failure load of radius at 12 months | 0.74 (8.3) | 0.09 (8.5)
  Change (%) from baseline in stiffness of tibia at 12 months | -0.01 (5.3) | 0.44 (5.0)
  Change (%) from baseline in failure load of tibia in 12 months | 0.08 (4.4) | 0.37 (4.4)
Statistical Analysis 1: Comparison: Testosterone Arm vs Placebo Arm; Test type: Superiority; p < 0.05, Kruskal-Wallis; Mean Difference (Final Values) = 3.6

2. Secondary Outcome: Markers of Bone Turnover to Measure Bone Metabolism
Description: Two markers of bone resorption, serum C-telopeptide (CTX) and tartrate-resistant acid phosphatase 5b (TRAP5b) and 2 markers of bone formation osteocalcin (OCN) and N-terminal propeptide of type 1 collagen (P1NP) will be evaluated. These markers will be obtained at months 0, 6, and 12. Enzyme-linked immunosorbent assay will be used to measure serum CTX (serum crosslaps, Osteometer, Hawthorne, CA), tartrate-resistant acid phosphatase 5b (TRAP5b) (EIA) (Microvue Bonehealth, Quidel Corporation, Biosource); and serum osteocalcin (ALPCO, Salem, NH). Serum P1NP will be measured by competitive radioimmunoassay (UniqTM P1NP RIA, Immunodiagnostic Systems, Scottsdale, AZ). Coefficients of variations for these assays are <10%.
Time Frame: months 0, 6 and 12
Measure: Mean (Standard Deviation); unit: % Change
Arm/Group | Testosterone Arm | Placebo Arm
Number analyzed (Participants) | 32 | 31
% Change
  Change (%) in osteocalcin from baseline at 6 months | -9.7 (47.5) | 17.4 (88.8)
  Change (%) in osteocalcin at 12 months | 7.8 (63) | 33.8 (87.5)
  Change (%) in C-telopeptide (CTX) from baseline at 6 months | -81.6 (10.6) | -80.4 (12.5)
  Change (%) in CTX from baseline at 12 months | 15.7 (64.2) | -1.4 (51.7)
  Change (%) in N-terminal peptide of type 1 collagen (P1NP) from baseline at 6 months | -8.6 (56.1) | -31.1 (34.5)
  Change (%) in P1NP from baseline at 12 months | 2.31 (60.2) | -23.1 (56.6)

3. Secondary Outcome: Osteoblast and Osteoclast Progenitor Cells Which Are Cells Found in Bone
Description: Osteoblast and osteoclast progenitor cells will be harvested from the serum at baseline, 6 and 12 months.
Time Frame: months 0, 6 and 12
Population: Out of the 44 participants who finished the study in testosterone arm, the cells did not stain in 3 patients. Out of the 42 participants who finished in the placebo, cells did not stain in one and the another was unable to provide enough blood sample for analysis at the end of the study
Measure: Mean (Standard Deviation); unit: % Change
Arm/Group | Testosterone Arm | Placebo Arm
Number analyzed (Participants) | 41 | 40
% Change
  Change (%) in osteoblast progenitor cells from baseline at 6 months | 5.1 (40.5) | -4.4 (36.9)
  Change (%) in osteoblast progenitor cells from baseline at 12 months | 10.8 (55.2) | -10.4 (29.5)
  Change (%) in osteoclast precursors from baseline at 6 months | 68.4 (161.6) | 19.2 (104.4)
  Change (%) in osteoclast precursors from baseline at 12 months | 59.1 (161.0) | 56.0 (130.1)

ADVERSE EVENTS:
Time Frame: Through study completion, i.e. approximately, 1 year.
Arm/Group | Testosterone Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 3/46 | 4/46
Other Adverse Events (participants affected / at risk) | 10/46 | 8/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Arm (N=46) | Placebo Arm (N=46)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphocytic leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting and constipation secondary to gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neuroendocrine tumor (Endocrine disorders) | 1 (1) | 0 (0)
Vomiting and bloody stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Arm (N=46) | Placebo Arm (N=46)
Pain and rashes at the site of drug application (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Anxious and having anger issues (Psychiatric disorders) | 1 (1) | 0 (0)
Trouble sleeping and mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Abscess on he right breast (Infections and infestations) | 1 (1) | 0 (0)
High prostate-specific antigen (Renal and urinary disorders) | 0 (0) | 2 (2)
High hematocrit (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fracture of greater trochanter after a fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
head trauma, rib pain and laceration of forehead after assault by the neighbor (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
C6-7 and rotator cuff surgeries from an injury sustained before he was enrolled in the study (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
C7-T1 disc injury from MVA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in the groin area after a car accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Outpatient knee surgery for meniscal tear. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar 4 vertebral fracture after picking-up a 375 lb. patients during an emergency (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left biceps tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Achilles tendon rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03887936/Prot_001.pdf
  • Statistical Analysis Plan (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03887936/SAP_002.pdf
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03887936/ICF_000.pdf